CLINICAL TRIAL: NCT04269330
Title: Comparison of Size Mesh and Undersized Mesh in Open Inguinal Hernia Repair: A Prospective, Randomized Study
Brief Title: Normal and Small Size Mesh in Open Inguinal Herni Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Alpaslan Şahin, Medical Doctor, principal investigator, General Surgery Department, Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Konya EAH
Record Dates: First submitted 2020-02-03; First posted 2020-02-13 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: General Surgery; Inguinal Hernia; Ventral Hernia
Keywords: mesh size; lichtenstein hernia repair; surgical technique
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-Normal size mesh in open inguinal herni (Sham Comparator): Comparison of normal and small size mesh in open inguinal hernia repair: Multicenter Prospective Randomized Controlled Trial.
  Interventions: Procedure: Comparison of normal and small size mesh in open inguinal hernia repair: Multicenter Prospective Randomized Controlled Trial.
- 2- small size mesh in open inguinal herni (Active Comparator): Comparison of normal and small size mesh in open inguinal hernia repair: Multicenter Prospective Randomized Controlled Trial.
  Interventions: Procedure: Comparison of normal and small size mesh in open inguinal hernia repair: Multicenter Prospective Randomized Controlled Trial.

INTERVENTIONS:
Procedure: Comparison of normal and small size mesh in open inguinal hernia repair: Multicenter Prospective Randomized Controlled Trial. — Comparison of normal and small size mesh in open inguinal hernia repair: Multicenter Prospective Randomized Controlled Trial.

SUMMARY:
Recent years, lots of treatment teqnique have development. We aimed that comparising the normal and small size meshes in the inguinal hernia patients.

DETAILED DESCRIPTION:
Data Collection Method: The research will be a multicentric, prospective and randomized clinical study to be conducted between 01.11.2018 and 28.02.2019 by the general surgery clinics of Mogadishu-Somalia Recep Tayyip Erdogan Training and Research Hospital and Health Sciences University Konya Training and Research Hospital.

Male patients with inguinal hernia repair will be included in the study. Patients will be randomized into two groups. While the normal size of 15 x 7 cm (105 cm2) mesh was used in the first group, In the second group, a small size 11 x 5 cm (55 cm2) mesh will be used.

Dismissal criteria are; Female patients, relapse hernias, bilateral inguinal hernia, laparoscopic hernia repair, diabetic patients using insulin, patients with COPD, peripheral vascular disease, emergency inguinal hernia repair, patients with high ASA score, patients with serious cardiological problems, heavy smokers, transfusions during the perioperative period.

Patients will be given clear and understandable information about the study. Patients who agree to participate in the study will receive a consent form explaining that they have participated in the study voluntarily.

Randomization is done by the secretary with a computer program. A note stating which group the patient is in is placed in a closed envelope and an envelope is opened at the preoperative surgery table.

The method of operation will be open inguinal hernia repair (Lichtenstein hernia repair). The patient will be repaired with mesh suitable for the randomization group. Operations will be performed under the supervision of an experienced surgeon or experienced surgeon.

Surgical Method: Patients will receive open inguinal hernia repair, known as Lichtenstein hernia repair. According to the Gilbert classification, the hernia type is recorded in the patient file.

Evaluation of patient characteristics and pain: the researcher will not know in which group the patients are. Demographic features, duration of surgery, hernia type, early postoperative complications, return to work will be recorded in the study forms. If there is a suspicion of recurrence in the physical examination, a recurrence assessment will be performed by ultrasonography and magnetic resonance examination if necessary. Recurrences will be detected at 1, 6, 12, and 24 and recorded on the study form.

Values will be recorded in the form by using the Sheffield Scale in the assessment of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* ages must be upper 18

Exclusion Criteria:

* Morbit obesity (BMI>40)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
The success of treatment. | 1 year
  The success of normal size mesh with small mesh as a result of hernia treatment

SECONDARY OUTCOMES:
patient satisfaction | 1 year
  As a result of hernia treatment, the patient's satisfaction in normal size mesh with small mesh is achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Alpaslan Şahin, MD, Principal Investigator — Konya Training and Research Hospital, Department of General Surgery
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

REFERENCES:
- [Background] Kulacoglu H, Celasin H, Oztuna D. Individual mesh size for open anterior inguinal hernia repair: an anthropometric study in Turkish male patients. Hernia. 2019 Dec;23(6):1229-1235. doi: 10.1007/s10029-019-01993-x. Epub 2019 Jun 20. PMID 31222460
- [Background] Anitha B, Aravindhan K, Sureshkumar S, Ali MS, Vijayakumar C, Palanivel C. The Ideal Size of Mesh for Open Inguinal Hernia Repair: A Morphometric Study in Patients with Inguinal Hernia. Cureus. 2018 May 3;10(5):e2573. doi: 10.7759/cureus.2573. PMID 29974028
- [Background] Seker D, Oztuna D, Kulacoglu H, Genc Y, Akcil M. Mesh size in Lichtenstein repair: a systematic review and meta-analysis to determine the importance of mesh size. Hernia. 2013 Apr;17(2):167-75. doi: 10.1007/s10029-012-1018-y. Epub 2012 Nov 11. PMID 23142904